CLINICAL TRIAL: NCT05245526
Title: Validate SpO2 Accuracy of Noninvasive Stryker Disposable Pulse Oximeter Sensors With Hypoxia at Rest
Brief Title: SpO2 Accuracy of Noninvasive Disposable Pulse Oximeter Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Sustainability Solutions (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRD10298
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Healthy; Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Healthy adult participants (Experimental): All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors.
  Interventions: Device: STRYKER SUSTAINABILITY SOLUTIONS PULSE OXIMETERS

INTERVENTIONS:
Device: STRYKER SUSTAINABILITY SOLUTIONS PULSE OXIMETERS — Reprocessed noninvasive pulse oximeter sensors.

SUMMARY:
The purpose of this clinical study is to validate the SpO2 accuracy of the Stryker Sustainability Solutions pulse oximetry sensors during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. The end goal is to provide supporting documentation for the SpO2 accuracy validation of the reprocessed sensors.

DETAILED DESCRIPTION:
In this study, the level of oxygen within the blood will be reduced in a controlled manner by reducing the concentration of oxygen the participant breathes. The accuracy of a noninvasive pulse oximeter sensor will be assessed by comparison to the oxygen saturation measurements from a laboratory blood gas analyzer.

It is required that the Accuracy Root Mean Square (ARMS) performance of the Stryker pulse oximetry sensors will meet a specification of +/-3% or better in non-motion conditions for the range of 70 - 100% SaO2 (typically, saturation is determined once with air breathing and then at one of 3 levels, e.g. 95%, 85%, and 75% saturation for about 30-60 seconds at each level), thereby demonstrating an acceptable SpO2 accuracy performance specification.

ELIGIBILITY:
Inclusion Criteria:

* Good general health with no evidence of pre-existing medical problems
* Fluent in both written and spoken English
* Must be able to review informed consent and is willing to comply with study procedures

Exclusion Criteria:

* Obesity (BMI >30)
* Known history of heart disease, lung disease, kidney or liver disease
* Prior diagnosis of asthma, sleep apnea, or use of CPAP
* Diabetes
* Clotting disorder
* Hemoglobinopathy or history of anemia that in the opinion of the investigators would make them unsuitable for study participation
* Any serious systemic illness
* Current smoker
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigator would interfere with the sensors working correctly
* History of fainting or vasovagal response
* History of sensitivity to local anesthesia
* Prior diagnosis of Raynaud's disease
* Unacceptable collateral circulation based on exam by investigators (Allen's test)
* Pregnant, lactating, or trying to get pregnant
* Unable or unwilling to provide informed consent, or unable or unwilling to comply with study procedures
* Any other condition which in the opinion of the investigators would make them unsuitable for the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Bickler, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Hypoxia Research Laboratory, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Data to be used by Sponsor only.

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adult Participants: All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors.
  STRYKER SUSTAINABILITY SOLUTIONS PULSE OXIMETERS: Reprocessed noninvasive pulse oximeter sensors.
  Device 1: Masimo RD Set Pulse Oximeter Sensor, 4000 Adt (non-woven butterfly style tape)
  Device 2: Masimo RD Set Pulse Oximeter Sensor, 4003 Neo (woven style tape)
Period: Overall Study
Arm/Group | Healthy Adult Participants
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Adult Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2
  Black or African American | 3
  Asian | 4
  Hispanic | 1
  Multiethnic | 2
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Percentage of SpO2 (oxygen saturation by pulse oximetry) measured by the Reprocessed Oximeter pulse oximetry sensors during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. Accuracy root mean square (ARMS) between measured SpO2 and reference SaO2 (arterial oxygen saturation) must meet the 3% specification for each reprocessed pulse oximetry sensor style. Accuracy will be determined by comparing the noninvasive blood oxygen saturation measurement of the pulse oximeter to that obtained from a blood sample and calculating the arithmetic root mean square error (Arms) value. Standard deviation of the differences is computed as the precision. Square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-2 hours
Measure: Number; unit: Root Mean Square Error (%)
Groups:
- Device 1: Reprocessed Masimo RD Set Pulse Oximeter Sensor, 4000 Adt; Device 2: Reprocessed Masimo RD Set Pulse Oximeter Sensor, 4003 Neo: All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors.
Arm/Group | Device 1: Reprocessed Masimo RD Set Pulse Oximeter Sensor, 4000 Adt | Device 2: Reprocessed Masimo RD Set Pulse Oximeter Sensor, 4003 Neo
Number analyzed (Participants) | 12 | 12
Root Mean Square Error (%) | 2.04 | 2.11

ADVERSE EVENTS:
Time Frame: 2 days
Groups:
- Device 1; Device 2: All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors.
Arm/Group | Device 1 | Device 2
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT05245526/Prot_SAP_000.pdf